CLINICAL TRIAL: NCT07306754
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Single Ascending Doses (SAD) of ABBV-243 in Healthy Adult Subjects and a Single Dose in Healthy Asian Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of ABBV-243 in Healthy Adults.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: M25-776
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1: ABBV-243 or Placebo (Experimental): Participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent, on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 2: ABBV-243 or Placebo (Experimental): Participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent, on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 3: ABBV-243 or Placebo (Experimental): Participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent, on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 4: ABBV-243 or Placebo (Experimental): Participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent. on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 5: ABBV-243 or Placebo (Experimental): Participants will receive either a single subcutaneous (SC) dose of ABBV-243, or the placebo equivalent, on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 6: ABBV-243 or Placebo (Experimental): Participants will receive either a single subcutaneous (SC) dose of ABBV-243, or the placebo equivalent, on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 7: ABBV-243 or Placebo (Experimental): Han Chinese participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent. on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo
- Group 8: ABBV-243 or Placebo (Experimental): Japanese participants will receive either a single intravenous (IV) dose of ABBV-243, or the placebo equivalent. on Day 1
  Interventions: Drug: ABBV-243; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-243 — Intravenous (IV) Infusion
  Arms: Group 1: ABBV-243 or Placebo; Group 2: ABBV-243 or Placebo; Group 3: ABBV-243 or Placebo; Group 4: ABBV-243 or Placebo; Group 7: ABBV-243 or Placebo; Group 8: ABBV-243 or Placebo
Drug: Placebo — Intravenous (IV) Infusion
  Arms: Group 1: ABBV-243 or Placebo; Group 2: ABBV-243 or Placebo; Group 3: ABBV-243 or Placebo; Group 4: ABBV-243 or Placebo; Group 7: ABBV-243 or Placebo; Group 8: ABBV-243 or Placebo
Drug: ABBV-243 — Subcutaneous (SC) Injection
  Arms: Group 5: ABBV-243 or Placebo; Group 6: ABBV-243 or Placebo
Drug: Placebo — Subcutaneous (SC) Injection
  Arms: Group 5: ABBV-243 or Placebo; Group 6: ABBV-243 or Placebo

SUMMARY:
The objective of this study is to assess the safety, tolerability, pharmacokinetics and immunogenicity of either single ascending intravenous (IV) doses of ABBV-243 or single ascending subcutaneous (SC) doses of ABBV-243 in healthy adult participants (Part 1), and a single intravenous (IV) dose in healthy Asian adult volunteers (Part 2

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 60 years of age inclusive at the time of Screening.
* BMI is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenth's decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Females, Non-Childbearing Potential are eligible as defined by meeting the following criteria:

  * Permanent sterility due to a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
  * Non-surgical permanent infertility due to Mullerian agenesis, androgen insensitivity, or gonadal dysgenesis; investigator discretion should be applied to determining study entry.
  * Postmenopausal female who is age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level ≥ 30 IU/L.
  * Postmenopausal female who is age > 55 years with no menses for 12 or more months without an alternative medical cause.
* Females, Childbearing Potential are defined as all other females who do not meet the above criteria and must adhere to the following:

  * Must not be pregnant or breastfeeding.
  * Must agree to avoid pregnancy while taking study treatment(s) and for at least 200 days after the last dose of study treatment.
  * Must agree to use a contraceptive method listed below (as per local regulations) that is highly effective (with a failure rate of < 1% per year, when used consistently and correctly). Participants must provide documentation to the site.
  * Bilateral tubal occlusion/ligation.
  * Intrauterine device (IUD) to be inserted at least 30 days prior to Screening.
  * Intrauterine hormone-releasing system (IUS) to be inserted at least 30 days prior to Screening.
* Part 2 only:

Healthy Japanese and Han Chinese male or female; between 18 and 60 years of age, inclusive at the time of Screening.

- Han Chinese participants must be first- or second-generation Han Chinese of full Chinese parentage. First-generation participants are defined as those born in China to two parents and four grandparents also born in China of full Chinese descent. Second-generation participants are defined as those born outside of China to two parents and four grandparents born in China of full Chinese descent.

OR

- Japanese participants must be first- or second-generation Japanese of full Japanese parentage. First-generation participants will have been born in Japan to two parents and four grandparents also born in Japan of full Japanese descent. Second-generation subjects born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent.

Exclusion Criteria:

* History: of epilepsy, any clinically significant cardiovascular, respiratory (except mild asthma as a child), renal, endocrine, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma, or localized carcinoma in situ of the cervix.
* History or evidence of active Tuberculosis (TB) disease or latent TB infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 204
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of ABBV-243 | Up to Day 204
  Maximum observed serum concentration (Cmax) of ABBV-243
Time to Cmax (Tmax) of ABBV-243 | Up to Day 204
  Time to Cmax (Tmax) of ABBV-243
Area Under the Serum Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUCt) of ABBV-243 | Up to Day 204
  Area under the serum concentration-time curve (AUC) from time 0 to the time of last measurable concentration (AUCt) of ABBV-243
Area Under the Serum Concentration-Time Curve From Time 0 to Infinite Time (AUCinf) of ABBV-243 | Up to Day 204
  AUC from time 0 to infinite time (AUCinf) of ABBV-243
Terminal Phase Elimination Rate Constant (β) of ABBV-243 | Up to Day 204
  Terminal phase elimination rate constant of ABBV-243
Terminal Phase Elimination Half-Life (t1/2) of ABBV-243 | Up to Day 204
  Terminal phase elimination half-life of ABBV-243
Anti-Drug Antibody (ADA) of ABBV-243 | Up to Day 204
  Confirmed Positive ADA Results.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 279789, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-776